CLINICAL TRIAL: NCT06822439
Title: Investigating the Acceptability and Feasibility of Remote Fetal Monitoring in a High Risk Obstetric Population
Brief Title: Remote Fetal Monitoring in High Risk Pregnancies
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Biorithm Pte Ltd (Industry)
Responsible Party: Principal Investigator, Ethan Litman, Clinical Fellow, Division of Maternal Fetal Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2024P000011
Record Dates: First submitted 2025-02-03; First posted 2025-02-12 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: High Risk Pregnancy; Remote Patient Monitoring; Diabetes; Hypertension
Keywords: Pregnancy; Non invasive testing; Remote patient monitoring
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Remote Monitoring: A cohort of patients with high risk pregnancies who will wear a remote monitoring device
  Interventions: Device: Fetal ECG monitoring

INTERVENTIONS:
Device: Fetal ECG monitoring — Patients will wear a fetal ECG monitor which they will place on their abdomen

SUMMARY:
Antenatal nonstress tests (NSTs) are performed to assess fetal health and are used as a cost-effective test that can be widely administered. However, an NST is operator-dependent due to the nature of Doppler ultrasound and is primarily performed in a clinic and hospital setting.

The ability to conduct a clinically valuable test at home would address access to care issues faced by numerous women in the United States and reduce the workload on healthcare clinicians facing a shortage of human resources.

This pilot study aims to assess the feasibility and acceptability of home NST monitoring in order to determine whether femomTM could be utilized as an adjunct to routine prenatal care.

Patients with high risk pregnancies who are recommended to undergo at least once weekly at 32 weeks testing by the obstetrician will be recruited for participation in this study. Participants will be asked to perform three 30 minute monitoring sessions weekly starting at 32 weeks for 6 weeks.

DETAILED DESCRIPTION:
Measuring fetal heart rate (FHR) through various methods is essential for assessing fetal wellbeing antenatally. This enables clinicians to identify patterns that could indicate fetal hypoxia.

Cardiotocography (CTG), which uses Doppler ultrasound, is the gold standard for non-invasive FHR monitoring. This technology detects movement in the cardiac structures and approximates the FHR from this and requires signal modulation and auto-correlation to provide accurate quality readings of FHR. This method of external FHR monitoring is prone to signal loss, maternal fetal ambiguity where the maternal heart rate is confused for FHR, and signal artefacts (e.g., double-counting, and half-counting), during both antenatal and intrapartum monitoring, and must be performed by an obstetric provider.

Non-invasive fetal electrocardiography (NIFECG) is a form of electrocardiography (ECG), which captures simultaneous maternal and fetal PQRST waves. NIFECG has the theoretical benefits of minimizing maternal-fetal heart activity confusion, is not affected by maternal adiposity, and delivers no energy to the patient, which permits prolonged periods of fetal monitoring with safety. To date, NIFECG has mostly been limited to research use due to low fetal signal-to-noise ratios. Despite technical challenges, NIFECG may be the most promising method of ambulatory self-applied FHR monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Intrauterine pregnancy greater than 32 weeks gestation
* Recommended for at least once weekly antenatal fetal testing by their obstetrician
* English-speaking

Exclusion Criteria:

* Under age 18 years of old
* Non-english speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High risk pregnancies that are recommend to undergo at least once weekly in-office antenatal testing.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent of sessions completed | 6 weeks
  Percentage of completed remote monitoring sessions
Percentage of interpretable sessions | 6 weeks
  Percentage of interpretable monitoring sesions

SECONDARY OUTCOMES:
Patient satisfaction | 6 weeks
  Patient satisfaction with device using a Likert rating scale (range 1 - 5)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study assessing the feasibility of using a novel device. We do not plan to share survey data from participants.